CLINICAL TRIAL: NCT03296930
Title: Effect Of Interferon-Free Direct Acting Antiviral Agents For Treatment Of Hepatitis C Virus Patients On The Normal Kidney
Brief Title: Effect Of DAAs For Treatment Of HCV On Normal Kidney
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hazem shoman, principle investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAAs on Normal Kidney
Record Dates: First submitted 2017-09-16; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Antiviral Drug Adverse Reaction
Keywords: Direct Acting Antiviral Agents (DAAs)
MeSH Terms: interventions — Sofosbuvir; Tablets; daclatasvir; Ribavirin; ombitasvir

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first drug group (Active Comparator): Sofosbuvir 400 MG Oral Tablet
  Interventions: Drug: Sofosbuvir 400 MG Oral Tablet,
- second drug group (Active Comparator): Ombitasvir/paritaprevir/ritonavir
  Interventions: Drug: Ombitasvir/paritaprevir/ritonavir

INTERVENTIONS:
Drug: Sofosbuvir 400 MG Oral Tablet, — Interferon free direct acting antiviral drugs used for treatment of HCV.
  Other Names: daclatasvir; ribavirin
  Arms: first drug group
Drug: Ombitasvir/paritaprevir/ritonavir — Interferon free direct acting antiviral drugs used for treatment of HCV.
  Other Names: ribavirin
  Arms: second drug group

SUMMARY:
The aim of the study is to determine the effect of different direct acting antiviral drugs used for treatment of chronic HCV infected patients on normal kidney.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a major health problem. The World Health Organization (WHO) estimated that at least 150-170 million people, approximately 3% of the world's population, are chronically infected. These patients are known to be at risk of developing liver complications, i.e., cirrhosis and liver cancer, with an estimated liver-related mortality of 350,000 people/year. However, the risks of morbidity and mortality are underestimated because they do not take into account the extra-hepatic consequences of HCV infection. Numerous extra-hepatic manifestations (HCV-EHMs) have been reported. In some large cohort studies, up to 74% of patients experienced HCV-EHMs of different severity, from perceived to disabling conditions.

Treatment of HCV infection has a long history. It began with interferon (IFN) mono-therapy, with less than 20% sustained virological response (SVR). Milestones include the addition of ribavirin (RBV) to the treatment protocol and providing pegylated-IFN (PegIFN) as an alternative treatment.

Treatment with PegIFN/RBV was the standard of care for about 10 years. The success rate of treatment with this regimen is very dependent on patient characteristics, including age, body mass index, ethnicity, and genetic factors.

Viral factors, especially HCV genotype, also affect the response to HCV treatment, and there are always additional factors that should be taken into account in each treatment approach, including treatment success rate, duration, cost, and side effects.

In light of these concerns, attempts have continued to introduce better therapeutic regimens.

Treatment of chronic HCV infection has been revolutionized in recent years. The FDA has approved different IFN-free direct acting antiviral regimens (DAAs) including: Sofosbuvir (SOF) in combination with Ledipasvir (LDV), combination of Ombitasvir/Paritaprevir/ Dasabuvir (a three direct acting antiviral, or 3D), combination therapy with Grazoprevir/Elbasvir (GZR/EBR), Simeprevir (SMV) and Daclatasvir (DCV) also in combination with SOF.

More than 95% of patients have a sustained viral response (SVR) using DAA. The recent Cohort studies have demonstrated that the new regimens of DAAs may be associated with renal side effects, especially when using SOF combinations. So, to aid in the correct use of DAAs in treatment of HCV patients, their potential renal toxicity must be known.

The close monitoring of renal function is required. Although, new DAAs were well tolerated, recent real-life studies have demonstrated some nephrotoxic effect in Frail populations treated with SOF based regimens.

The use of direct acting antiviral agents (DAAs) in HCV patients might be expected to result in improved outcomes in hepatic functions even in end stage liver disease. But, the effect of DAAs on the kidney still needing a specific study.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients with age above 18 years presented with chronic HCV infection (diagnosed by HCV RNA positive) with normal kidney functions, i.e.:

  * Normal S.creatinine
  * Normal urine analysis (without proteinuria, haematuria or abnormal casts).
  * Normal renal sonography.
* and candidate for direct acting antiviral drugs.

Exclusion Criteria:

* Any chronic HCV patient with known renal disease.
* Patients with abnormal kidney functions, i.e.:

  * Abnormal S.creatinine.
  * Abnormal urine analysis (with proteinuria, haematuria or abnormal casts).
  * Abnormal renal US
* Any other known renal disease (lupus nephritis, diabetic nephropathy).
* Severe co-morbidity as severe heart failure or malignancy.
* Other liver disease (autoimmune hepatitis, HBV, Wilson, ……).
* Decompansated liver disease (ascites, hepatic encephalopathy, …).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Effect of the direct acting antiviral agents used for HCV treatment on the function of the normal kidney by measurement of serum creatinine. | one year
  assessment of the renal toxicity of direct acting antivirals used for HCV treatment by measurement of the serum creatinine to detect any deviation beyond the normal values.

CONTACTS AND LOCATIONS:
Overall Officials: Zainelabdeen A Sayed, MD, Study Chair — Assistant Professor of Internal Medicine; Mohammed M Abdallah, MD, Study Chair — Professor of Internal Medicine

REFERENCES:
- [Background] Behnava B, Sharafi H, Keshvari M, Pouryasin A, Mehrnoush L, Salimi S, Karimi Elizee P, Ghazimoghaddam M, Alavian SM. The Role of Polymorphisms Near the IL28B Gene on Response to Peg-Interferon and Ribavirin in Thalassemic Patients With Hepatitis C. Hepat Mon. 2016 Jan 23;16(1):e32703. doi: 10.5812/hepatmon.32703. eCollection 2016 Jan. PMID 27110259
- [Background] Cacoub P, Gragnani L, Comarmond C, Zignego AL. Extrahepatic manifestations of chronic hepatitis C virus infection. Dig Liver Dis. 2014 Dec 15;46 Suppl 5:S165-73. doi: 10.1016/j.dld.2014.10.005. Epub 2014 Nov 8. PMID 25458776
- [Background] Carrier P, Essig M, Debette-Gratien M, Sautereau D, Rousseau A, Marquet P, Jacques J, Loustaud-Ratti V. Anti-hepatitis C virus drugs and kidney. World J Hepatol. 2016 Nov 18;8(32):1343-1353. doi: 10.4254/wjh.v8.i32.1343. PMID 27917261
- [Background] European Association for Study of Liver. EASL Recommendations on Treatment of Hepatitis C 2015. J Hepatol. 2015 Jul;63(1):199-236. doi: 10.1016/j.jhep.2015.03.025. Epub 2015 Apr 21. No abstract available. PMID 25911336
- [Background] Ferenci P, Bernstein D, Lalezari J, Cohen D, Luo Y, Cooper C, Tam E, Marinho RT, Tsai N, Nyberg A, Box TD, Younes Z, Enayati P, Green S, Baruch Y, Bhandari BR, Caruntu FA, Sepe T, Chulanov V, Janczewska E, Rizzardini G, Gervain J, Planas R, Moreno C, Hassanein T, Xie W, King M, Podsadecki T, Reddy KR; PEARL-III Study; PEARL-IV Study. ABT-450/r-ombitasvir and dasabuvir with or without ribavirin for HCV. N Engl J Med. 2014 May 22;370(21):1983-92. doi: 10.1056/NEJMoa1402338. Epub 2014 May 4. PMID 24795200
- [Background] Haj-Sheykholeslami A, Keshvari M, Sharafi H, Pouryasin A, Hemmati K, Mohammadzadehparjikolaei F. Interferon-lambda polymorphisms and response to pegylated interferon in Iranian hepatitis C patients. World J Gastroenterol. 2015 Aug 7;21(29):8935-42. doi: 10.3748/wjg.v21.i29.8935. PMID 26269684
- [Background] Kwo P, Gitlin N, Nahass R, Bernstein D, Etzkorn K, Rojter S, Schiff E, Davis M, Ruane P, Younes Z, Kalmeijer R, Sinha R, Peeters M, Lenz O, Fevery B, De La Rosa G, Scott J, Witek J. Simeprevir plus sofosbuvir (12 and 8 weeks) in hepatitis C virus genotype 1-infected patients without cirrhosis: OPTIMIST-1, a phase 3, randomized study. Hepatology. 2016 Aug;64(2):370-80. doi: 10.1002/hep.28467. Epub 2016 Mar 22. PMID 26799692
- [Background] Lee SS, Bain VG, Peltekian K, Krajden M, Yoshida EM, Deschenes M, Heathcote J, Bailey RJ, Simonyi S, Sherman M; CANADIAN PEGASYS STUDY GROUP. Treating chronic hepatitis C with pegylated interferon alfa-2a (40 KD) and ribavirin in clinical practice. Aliment Pharmacol Ther. 2006 Feb 1;23(3):397-408. doi: 10.1111/j.1365-2036.2006.02748.x. PMID 16422999
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Pawlotsky JM. New hepatitis C therapies: the toolbox, strategies, and challenges. Gastroenterology. 2014 May;146(5):1176-92. doi: 10.1053/j.gastro.2014.03.003. Epub 2014 Mar 12. PMID 24631495
- [Background] Sharafi H, Alavian SM. IL28B polymorphism, Explanation for Different Responses to Therapy in Hepatitis C Patients. Hepat Mon. 2011 Dec;11(12):958-9. doi: 10.5812/kowsar.1735143X.794. Epub 2011 Dec 20. No abstract available. PMID 22368678
- [Background] Sulkowski MS, Gardiner DF, Rodriguez-Torres M, Reddy KR, Hassanein T, Jacobson I, Lawitz E, Lok AS, Hinestrosa F, Thuluvath PJ, Schwartz H, Nelson DR, Everson GT, Eley T, Wind-Rotolo M, Huang SP, Gao M, Hernandez D, McPhee F, Sherman D, Hindes R, Symonds W, Pasquinelli C, Grasela DM; AI444040 Study Group. Daclatasvir plus sofosbuvir for previously treated or untreated chronic HCV infection. N Engl J Med. 2014 Jan 16;370(3):211-21. doi: 10.1056/NEJMoa1306218. PMID 24428467
- [Background] Tong MJ, Reddy KR, Lee WM, Pockros PJ, Hoefs JC, Keeffe EB, Hollinger FB, Hathcote EJ, White H, Foust RT, Jensen DM, Krawitt EL, Fromm H, Black M, Blatt LM, Klein M, Lubina J. Treatment of chronic hepatitis C with consensus interferon: a multicenter, randomized, controlled trial. Consensus Interferon Study Group. Hepatology. 1997 Sep;26(3):747-54. doi: 10.1002/hep.510260330. PMID 9303508
- [Background] Zeuzem S, Ghalib R, Reddy KR, Pockros PJ, Ben Ari Z, Zhao Y, Brown DD, Wan S, DiNubile MJ, Nguyen BY, Robertson MN, Wahl J, Barr E, Butterton JR. Grazoprevir-Elbasvir Combination Therapy for Treatment-Naive Cirrhotic and Noncirrhotic Patients With Chronic Hepatitis C Virus Genotype 1, 4, or 6 Infection: A Randomized Trial. Ann Intern Med. 2015 Jul 7;163(1):1-13. doi: 10.7326/M15-0785. PMID 25909356